CLINICAL TRIAL: NCT03086031
Title: A Randomised Controlled Trial of a Manual-Based Vocational Rehabilitation Program for Patients With Acquired Brain Injury
Brief Title: Manual-Based Vocational Rehabilitation Program for Patients With Acquired Brain Injury
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Brain Injury Center BOMI, Roskilde, Denmark (Other)
Collaborators: University of Copenhagen (Other); Rigshospitalet, Denmark (Other); Hospital de Cruces (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: 2016-41-4950
Record Dates: First submitted 2017-03-02; First posted 2017-03-22 (Actual); Last update posted 2017-07-13 (Actual); Status verified 2017-07

CONDITIONS: Brain Injuries
Keywords: Traumatic brain injury, Vocational rehabilitation, Caregiver intervention,
MeSH Terms: conditions — Brain Injuries; Brain Injuries, Traumatic

STUDY DESIGN:
Intervention Model Description: In order to avoid confounding between the VR intervention and the control group due to random probability, the number of cases and controls within each of the four municipalities is fixed to be the same (+1/-1). Due to the prospective nature of the inclusion, which practically means that the number of patients included within each municipality is not a priori known, the randomization is performed by randomly assigning the first patient within each municipality to either the VR intervention or the conventional VR program. The following patient (within each municipality) is then assigned consecutive to the other group and so forth. This randomization scheme ensures equal distribution of cases and controls both within each municipality as well as in time avoiding confounding by these two factors.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Due to the nature of the study, it is not possible to blind neither the participants nor the rehabilitation team, but they will be asked not to disclose any details about the allocation, or the content of the VR. The two independent research assistants will be trained to administer the assessments and will be blinded to the allocation when entering data into the database. The researchers and the statistician performing the data analysis are blind to the treatment arm in which the participants are allocated. The rehabilitation team and the research assistants will only be involved in the data collection and will therefore not participate in the data analyses.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Program-based vocational rehabilitation (Experimental): Combined intervention with a neuropsychological, social and community intervention followed by a vocational rehabilitation programme with a total length of 6-9 months.
  Interventions: Behavioral: Program -based vocational rehabilitation intervention
- Conventional vocational rehabilitation(controls) (Active Comparator): Individuals allocated to the control group will receive the conventional VR program provided by the four municipalities over the same period of time. Thus, the participants in the control group will receive VR support by the local municipal authority that may vary in content and intensity. As for the intervention group, each individual in the control group will select a family caregiver that will go through the same questionnaires as the caregivers in the VR intervention group regarding health-related quality of life and functional level. Furthermore, the case manager at the municipalities will oblige to (1) hand out the baseline questionnaires to the participants and their family caregivers, (2) complete a questionnaire about each participants at the beginning, the end of the study, and again at 6-month of follow-up.
  Interventions: Behavioral: Conventional vocational rehabilitation (controls)

INTERVENTIONS:
Behavioral: Program -based vocational rehabilitation intervention — The VR intervention lasts for a total of 6-9 months with first six different modules (3-month) that are individually planned, and second a work placement program (approximately 3-6 months). Each of the different modules follows a comprehensive "standard operating procedures" (SOP's). The six modules will be grouped into (a) individual therapies which includes neuropsychological sessions (10-hours), balance between work and everyday life (20-hours), and job matching (10-hours), (b) grouped-based therapies which includes psycho education (18-hours), mindfulness (15-hours), and physiotherapy training (15-hours), (c) an manualized family intervention program (8 sessions of 90 minutes), and an individual caregiver coaching (12-hours), (d) a work placement program including work practice (3-6 month), supported employment by the rehabilitation team (30-hours), and the development of a post rehabilitation plan (4-hours).
  Arms: Program-based vocational rehabilitation
Behavioral: Conventional vocational rehabilitation (controls) — Treatment as usual delivered by the municipalities.
  Arms: Conventional vocational rehabilitation(controls)

SUMMARY:
An acquired brain injury (ABI) is a complex injury often followed by a broad range of cognitive, physical, emotional, and behavioral disabilities. Because of these disabilities, vocational rehabilitation (VR) is a challenging task, however, of great importance, since approximately 75% of the patients with ABI are of working age. Thus, standardized clinically effective and cost-effective methodologies regarding VR for patients with ABI are highly needed.

This study is an interventional, two-arm, 6-month follow-up, cluster randomized controlled trial involving four municipalities in the Zealand Region and the Capital Region of Denmark. A total of 84 patients with ABI evenly distributed across four municipalities will be included in the study. The patients will randomly be allocated in a 1:1 ratio to the VR intervention provided by a specialized Brain Injury Centre or the conventional VR provided by the municipalities (usual care). The 6-9 month intervention will consist of individual and group therapies as well as a work placement program including supported employment. Furthermore, the intervention will include a family intervention program followed up by support to one individual family caregiver. The primary outcomes are increased work or study rate at 6-month follow-up. Moreover, a budget impact analysis and possibly a cost utility analysis of the intervention will be performed The program is one of the first to include a comprehensive and target VR intervention including multiple parties such as the municipalities, a specialized rehabilitation team, and patients' own family caregivers. If this intervention is proven successful when compared to the conventional VR, it will provide evidence for a manual-based individualized holistic approach in returning to work after an ABI.

The first hypothesis of the study is that more participants allocated to the VR intervention group will have a significant higher employment/study rate (measured in hours) at 6-month follow-up when compared to participants receiving the conventional VR program provided by the municipalities (control group). The second hypothesis is that health-related quality of life (HRQoL) and disability among the participants as well as the HRQoL and caregiver burden among the caregivers are significantly improved at the end of the VR intervention and at 6-month follow-up when compared to the conventional VR program. Finally, a budget impact and possibly a cost utility analysis will be performed.

DETAILED DESCRIPTION:
An acquired brain injury (ABI) is a complex injury often followed by a broad range of cognitive, physical, emotional, and behavioral disabilities. Because of these disabilities, most patients with ABI find it challenging to remain in or return to work/education post-injury even though approximately 75% of these patients are of working age.

Vocational rehabilitation (VR) is often a prolonged process leading to high cost to the health care system and society. Barriers to VR success include the severity of the ABI, age at injury, income and education pre-injury, but also challenges directly related to the workplace. Often, the employer has little or no knowledge about the consequences of an ABI and, in addition, lack of communication regarding the challenges and needs in relation to work-related tasks influence the VR.

Even though returning to work has proven important for long term ABI survival and increased levels of quality of life standardized research-based VR programs targeting patents with ABI have been lacking. It has previously been shown that support from specialized VR teams help patients with ABI returning to work post-injury but only few studies have examined the long term effect.

Previous VR interventions have been performed similarly to all patients even though ABI is a broad diagnostic category with various degrees and characteristics. Thus, VR interventions that are tailored to each patient might be proven more efficient and effective in enhancing returning to work.

This study is an interventional, two-arm, 6-month follow-up, cluster randomized controlled trail including 84 participants with an ABI allocated randomly (allocation ratio 1:1) to the VR intervention and control group that consists of a conventional VR program (usual care).

The main objective of the study is to develop an individually targeted manual-based VR program and determine its efficacy for patients with ABI. It is hypothesized that

* more participants allocated to the VR intervention group will have a significant higher employment or study rate (measured in hours) at 6-month follow-up when compared to participants receiving the conventional VR program provided by the municipalities (control group).
* health-related quality of life (HRQoL) and disability among the participants and that HRQoL and caregiver burden among the caregivers are significantly improved at the end of the VR intervention and at 6-month follow-up when compared to the conventional VR program.

A budget impact and possibly a cost utility analysis will be performed since the investigators hypothesize that it will be an economically sound decision for the municipalities to invest in a specialized VR when compared to the conventional VR program.

The duration of the study is three years and the assessments will take place at baseline and at the end of the intervention (approximately after 6-9 months). In order to determine any long term effect of the intervention, follow-up assessment is planned after 6 months.

The 84 patients included in the study will be recruited from four municipalities in the Zealand Region and Capital Region of Denmark in the period between April 2017 and July 2017.

In order to avoid confounding between the VR intervention and the control group due to random probability, the number of cases and controls within each of the four municipalities is fixed to be the same (+1/-1). Due to the prospective nature of the inclusion, which practically means that the number of patients included within each municipality is not a priori known, the randomization is performed by randomly assigning the first patient within each municipality to either the VR intervention or the conventional VR program. The following patient (within each municipality) is then assigned consecutive to the other group.

This manual-based VR study comprises the following three phases:

1. Initial assessment: Within two weeks after the referral to the study, each patient will meet with the rehabilitation team of the project at the Brain Injury Centre BOMI (Roskilde, Denmark).The participant will be fully informed about the content of the study, how participation is voluntary, and how they are free to withdraw at any time during the study. If written informed consent is obtained, each patient are assigned a unique trial ID number and baseline questionnaires will be filled out together with the following socio-demographic, employment, and clinical data (gender, date of birth, residence, civil status, nationality, income, pre-injury employment and education status, pre-injury occupation status, length of education, time since the brain injury, type and location of the brain injury, number of days hospitalized, the date of discharge, clinical diagnoses or any relevant medical events, and alcohol consumption or abuse).

   Each patients included in the VR intervention group will be asked to choose at least two family members to participate in the family intervention and one family caregiver which will participate actively in the individual sessions and serve as future support and resource facilitator to assist them in returning to work.

   To exclude recruitment biases, patients that meet the eligibility criteria but refuse to participate in the study will be asked a few questions about their refusal.
2. The VR intervention program: The VR intervention lasts for a total of 6-9 months and consists of first six different modules (3-month) that are individually planned based on the patient needs and goals, and second a work placement program (approximately 3-6 month). To ensure a uniform procedure of each of the different modules, comprehensive "standard operating procedures" (SOP's) will be developed by the rehabilitation team at the Brain Injury Centre before the beginning of the VR intervention. All members of the rehabilitation team will be thoroughly trained in the VR intervention.

   The six modules will be grouped into (a) individual therapies which includes neuropsychological sessions (10-hours), balance between work and everyday life (20-hours), and job matching (10-hours), (b) grouped-based therapies which includes psycho education (18-hours), mindfulness (15-hours), and physiotherapy training (15-hours), (c) an manualized family intervention program (8 sessions of 90 minutes), and an individual caregiver coaching, supporting the caregiver in assisting the patient using the different strategies and tools learned in the intervention in everyday life and at the workplace (12-hours), (d) a work placement program including work practice (3-6 month), supported employment by the rehabilitation team (30-hours), and the development of a post rehabilitation plan (4-hours).
3. Post-trial evaluation: An evaluation of the VR intervention will be performed by a self-developed semi-structured interview of each patient. Here, questions related to the recruitment procedure, the modules of the study, the timing of modules, and the coaching by the rehabilitation team will be collected. Furthermore, will all case managers at the four municipalities that referred participants to the study be asked about their experiences.

Individuals allocated to the control group will receive the conventional VR program provided by the four municipalities over the same period of time. Thus, the participants in the control group will receive VR support by the local municipal authority that may vary in content and intensity. As for the intervention group, each individual in the control group will select a family caregiver that will go through the same questionnaires as the caregivers in the VR intervention group regarding health-related quality of life and functional level. Furthermore, the case manager at the municipalities will oblige to (1) hand out the baseline questionnaires to the participants and their family caregivers, (2) complete a questionnaire about each participants at the beginning, the end of the study, and again at 6-month of follow-up.

A budget impact analysis of the financial streams related to ABI for the two compared interventions will be performed to examine the affordability of the interventions. The health gains will be quantified by the standardized questionnaire EQ-5D-3L (health profiles, and self-perceived health status). If relevant and feasible, a cost-utility analysis (quality adjusted life years (QALYs)) from a societal perspective will be performed.

Data on financial streams and costs are collected from the patients when discharged from hospital to the end of the follow-up period of the study by a self-developed questionnaire to the participating municipalities. In order to calculate the present value of the future gains of the interventions a discount rate of 4 % will be applied. Statistical uncertainty on the results will be calculated, in addition, to sensitivity analysis on critical assumptions (difference-in-difference analysis).

Data will be stored in a secure password-protected electronic database hosted by the Brain Injury Centre BOMI following Danish legislation. Data will be collected prior to the intervention (baseline), after four months of intervention (month 4), at the end of the intervention (month 9), and a 6-month follow-up (month 15) by various questionnaires. All assessments will take place at the local rehabilitation center and will be done by 2-3 research assistants blinded to the intervention. Each assistant will receive thoroughly training in the assessment and will continue to be supervised throughout the study period

Ethical issues:

The study has been reported to the Danish Data Protection Agency (registration number 2016-41-4950). The Regional Ethical Committee of Copenhagen, Denmark, has stated that the study does not need their approval (komitélovens §1 and 2). The study will be carried out according to the local legal and regulatory requirements, and data will be handled according to the guidelines given by the Danish Personal Data Protection Agency.

All participants must give written and oral informed consent to participate in the study, including their consent to publish the results. If any participants are under the age of 18 they will provide a verbal acceptance while their parents will complete the written consent.

We expect a very low risk for adverse effects. However, increased fatigue in the intervention group could occur since a more intense program is followed. Furthermore, VR could for some participants be perceived as stressful and inclusion of the family caregivers could result in a higher risk for intra-family conflicts. The first session in the family intervention program includes psychoeducation in how to recognize, handle, and cope with situations that might escalate emotionally. All adverse effects will be reported.

Sample size and power:

The primary endpoint "hours at work/study per week" is assumed to follow a poisson distribution with an overdispersion of 4. Under this assumption, the relation between average hours at work for the conventional VR treatment, the expected surplus of hours by the VR intervention and the study power is calculated for a study with n = 42+42 = 84 participants. A study with 10 hours of work for the conventional VR treatment and 14 hours of work for the VR intervention leads to a study power of 0.8 at level alpha = 0.05.

Statistical analysis:

Baseline characteristics of the participants will be reported to ensure homogeneity between the VR intervention and the control group. Differences between baseline characteristics for continuous variables will be tested by an independent samples t-test /Mann-Whitney U test dependent on the distribution of the data. Categorical variables will be analyzed by a Chi-square test.

The differences between the VR intervention and the control group for the primary and secondary outcomes will be analyzed using repeated measurements statistical tools and multilevel analysis including possible confounders.

ELIGIBILITY:
Inclusion Criteria:

* suffers from an acquired brain injury
* acquired the brain injury within the last 3 to 24 months
* currently unemployed, but employed/enrolled at an education prior to the injury
* motivated to participate in vocational rehabilitation
* able to participate in group sessions
* able to understand and speak Danish
* have at least two Family caregivers willing to participate in the study

Exclusion Criteria:

* have any other somatic or psychiatric illnesses before the acquired brain injury that make it impossible to complete the intervention
* suffer from substance abuse or severe aphasia
* have a progressive brain injury
* are pregnant,
* have a mini mental state examination score <23.

Ages: 16 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 84 (Estimated)
Dates: Start 2017-08 (Estimated); Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Increased work/study rate at 6-month follow-up | Measurement assessed at baseline, and after 4 months, 9 months, and 15 months.
  The information will be recorded from the involved municipalities own registers and by interviews.

SECONDARY OUTCOMES:
Proficiency on functional task and functional status | Measurement assessed at baseline, and after 4 months, 9 months, and 15 months.
  Proficiency on functional task and functional status will be measured with The Mayo-Portland Adaptability Inventory (MPAI-4) and Glasgow Outcome Scale Extended
Health related quality of life | Measurement assessed at baseline, and after 4, 9 months and 15 months.
  Health related quality of life would be measured with EuroQol five dimensions questionnaire EQ-5D-3L which measures quality of life in five dimensions (mobility, self-care, usual activities, pain/discomfort, anxiety/depression) with three statements in each domain coded 1,2, or 3.
Anxiety and depression | Measurement assessed at baseline, and after 9 and 15 months.
  Hospital Anxiety and Depression Scale (HADS) scale are used to measure the symptoms of anxiety and depression in the patients. The final scale has a total of 14 items, with responses being scored on a scale of 0-3 (3 indicates higher symptom frequencies. Scores for each subscale (anxiety and depression) range from 0 to 21 with scores categorized as follows: normal 0-7, mild 8-10, moderate 11-14, and severe 15-21. Scores for the entire scale (emotional distress) range from 0 to 42.
Fatigue | Measurement assessed at baseline, and after 4, 9 and 15 months.
  The Dutch multifactor Fatigue Scale (DMFS) measures different aspects of fatigue after acquired brain injury. It consists of five dimensions ( 1:Mental fatigue, 2.Physical fatigue, 3.Impact of fatigue, 4.Signs and consequences and 5.Coping with fatigue). It has five subscale scores and no total score.
Physical function | Measurement assessed at baseline, and after 4 and 15 months.
  The Timed Up and Go (TUG) assess mobility by measuring the time (in seconds) used by the patient to walk a line of three meter, turn around and go back again.
Daily activity | Measurement assessed at baseline, and after 9 and 15 months.
  The Worker Role Interview (WRI) is a semi-structured interview designed to be used as the psychosocial/environmental component of the initial rehabilitation assessment process for the injured worker or the worker with a long term disability and poor/limited work history.
Problem Solving Inventory | Measurement assessed at baseline, and after 4 and 15 months.
  The Problem Solving Inventory (PSI) assesses perceptions of the patients problem-solving ability and behaviours and attitudes Associated with problem-solving style. The PSI consists of 35 items with a 6-point Likert scale (1=strongly agree to 6=strongly disagree).
Selv-perceived burden to others | Measurement assessed at baseline, and after 4,9 and 15 months.
  The Self-perceived Burden Scale (SPB) consists of 25 items rated on a five-point scale (1="none of the time" to 5="all of the time).
Executive functions | Measurement assessed at baseline, and after 4 and 15 months.
  TRAIL A and B. The Trail Making Test is a neuropsychological test of visual attention and task switching. It consists of two parts in which the subject is instructed to connect a set of 25 dots as quickly as possible while still maintaining accuracy.The test can provide information about visual search speed, scanning, speed of processing, mental flexibility, as well as executive functioning.
Perceived Stress | Measurement assessed at baseline, and after 4, 9 and 15 months.
  The Perceived Stress Scale (PSS) is a 10-item self-report measurement of stress with scores ranging from 0-4 and a maximum total score of 40.

OTHER OUTCOMES:
Outcome among Family caregivers (Quality of life). | Measurement assessed at baseline, and after 4 and 15 months.
  EuroQol five dimensions questionnaire EQ-5D-3L; questionnaire EQ-5D-3L which measures quality of life in five dimensions (mobility, self-care, usual activities, pain/discomfort, anxiety/depression) with three statements in each domain coded 1,2, or 3.
Adaptability and cohesion in the Family towards their new situation with a brain injured Family member. | Measurement assessed at baseline, and after 4 and 15 months.
  The Family Adaptability and Cohesion Scale (FACES-IV) assess Family cohesion and Family flexibility. It consists of 62 items.
Problem Solving Inventory among caregivers | Measurement assessed at baseline, and after 4 and 15 months.
  The Problem Solving Inventory (PSI) assesses perceptions of the problem-solving ability and behaviours and attitudes associated with problem-solving style. The PSI consists of 35 items with a 6-point Likert scale (1=strongly agree to 6=strongly disagree).
Burden among caregivers | Measurement assessed at baseline, and after 4 and 15 months.
  The caregiver burden scale (CBS) is a 22-item self-report Measurement that assess the felt burden among caregiver in taking care of their relatives. The items are scored on a five point likert scale ranging from never (0) to nearly always (4). The the total score is calculated with a total score of 0 to 20 (little or no burden), 21 to 40 (mild to moderate burden), 41 to 60 (moderate to severe burden) and 61 to 88 (severe burden).

CONTACTS AND LOCATIONS:
Overall Officials: Kirsten krogh Jensen, MBA, Study Director — Brain Injury Center BOMI

IPD SHARING:
Plan to Share IPD: Undecided
The identified individual participant data for all primary and secondary outcome measures might be interesting in follow-up analyses or in case-reports depending on the results of the study.

REFERENCES:
- [Derived] Hoeffding LK, Nielsen MH, Rasmussen MA, Norup A, Arango-Lasprilla JC, Kjaer UK, Burgdorf KS, Quas KJ, Schow T. A manual-based vocational rehabilitation program for patients with an acquired brain injury: study protocol of a pragmatic randomized controlled trial (RCT). Trials. 2017 Aug 10;18(1):371. doi: 10.1186/s13063-017-2115-0. PMID 28793916